CLINICAL TRIAL: NCT02320747
Title: Immediate Effect of Tai Chi Exercise in Healthy Volunteers:Randomized Controlled Study
Brief Title: Immediate Effect of Tai Chi Exercise in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adwin Life Care (Industry)
Collaborators: Shanghai University of Sport (Other); Warwick Research Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: Adwin009
Record Dates: First submitted 2014-12-10; First posted 2014-12-19 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Healthy
Keywords: Volunteers
MeSH Terms: interventions — Tai Ji

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tai Chi Group (Experimental): Experienced instructor at teaching tai chi delivered in a group setting in the community lasted approximately 40 minutes. Participants in the program served as an active control group that matched to the program and delivered.The class comprised mainly seated exercises including stretching, low-level strength, and low-level cardiovascular exercise. Participants walked (warm-up and cool-down) for 7 min in class, remaining seated or standing with arm support the rest of the time.
  Interventions: Other: Tai Chi
- Control Group (No Intervention)

INTERVENTIONS:
Other: Tai Chi
  Arms: Tai Chi Group

SUMMARY:
Tai Chi has been widely practiced as a Chinese martial art that focuses on slow sequential movements, providing a smooth, continuous and low intensity activity. It has been promoted to improve balance and strength and to reduce falls in the elderly, especially those 'at risk'. The potential benefits in healthy younger age cohorts and for wider aspects of health have received less attention.

The present study documented prospective changes in balance and vascular responses for a community sample of adults.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 25 years old
* Have given written informed consent
* Have a high school level of education
* Be healthy and psychologically stable as determined by screening for medical and psychiatric problems via a personal interview, a medical questionnaire, a physical examination, an electrocardiogram (ECG), and routine medical blood and urinalysis laboratory tests.
* Have an active interest in exploring and developing their spiritual lives
* Cigarette smokers must agree to abstain from smoking on session days
* Agree to refrain from using any psychoactive drugs, including alcoholic beverages, within 24 hours
* Agree that for one week before each session, refrain from taking any nonprescription medication, nutritional supplement, or herbal supplement except when approved by the study investigators.

Exclusion Criteria:

* Women who are pregnant or nursing
* Cardiovascular conditions: coronary artery disease, stroke, angina, uncontrolled hypertension, a clinically significant ECG abnormality
* Epilepsy with history of seizures
* Insulin-dependent diabetes
* Currently taking psychoactive prescription medication on a regular (e.g., daily) basis

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2014-09; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Heart rate (HR) | 40 Minutes
  Heart rate was recorded before and after the session.
Systolic Pressure (SP) | 40 minutes
Diastolic Pressure (DP) | 40 Minutes

CONTACTS AND LOCATIONS:
Overall Officials: Avinash Mishra, MSc, Principal Investigator — Shanghai University of Sport; Dinghai Yu, Study Director — Shanghai University of Sport
Locations (1):
- GyanSanjeevani, Jaipur, Rajasthan, India